CLINICAL TRIAL: NCT02259361
Title: Efficacy of Sustained-release Oral Dalfampridine on Upper Extremity Function in Patients With Multiple Sclerosis: a Pilot Study
Brief Title: Efficacy of Dalfampridine on Upper Extremity Function in Patients With MS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHEBA-13-0380-AA-CTIL
Record Dates: First submitted 2014-10-01; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — 4-Aminopyridine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Active Comparator): Intervention: Sustained-release oral dalfampridine, one 10 mg tablet, twice daily, taken 12 hours apart (one tablet in the morning and one tablet in the evening) for 14 consecutive days.
  Interventions: Drug: Sustained-release oral dalfampridine
- Placebo (Placebo Comparator): Placebo, one 10 mg tablet, twice daily, taken 12 hours apart (one tablet in the morning and one tablet in the evening) for 14 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sustained-release oral dalfampridine — One Sustained-release oral dalfampridine; 10 mg tablet, twice daily, taken 12 hours apart (one tablet in the morning and one tablet in the evening) taken for 14 consecutive days.
  Other Names: Prolonged-release Fampridine; Ampyra
  Arms: Experimental
Drug: Placebo — Placebo, 10 mg tablet, twice daily, taken 12 hours apart (one tablet in the morning and one tablet in the evening) taken for 14 consecutive days.
  Other Names: Active comparator
  Arms: Placebo

SUMMARY:
This study evaluates the effects of sustained-release oral dalfampridine in the treatment of upper limb deficits in people with multiple sclerosis (MS). In this double-blind randomized pilot study half of participants will dalfampridine, while the other half will receive a placebo.

DETAILED DESCRIPTION:
Dalfampridine (ampyra), a drug with a mechanism for symptomatic management of MS among blocks potassium channels on demyelinated neurons, allows normal electrical conduction.

Dalfampridine has recently been found to be associated with improvements in visual function, strength, ambulation, fatigue, and endurance in individuals with MS.

Although this medication has a widespread effect, its influence on upper extremity function has never been investigated in a double blind randomized case control study.

Following the fact that during the disease course, approximately 3 out of 4 multiple sclerosis patients encounter upper limb dysfunction the primary objective of this study will be to investigate the efficacy of sustained-release oral dalfampridine on upper extremity function in patients with MS.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have the ability to understand the purpose and risks of the study provide a signed and dated informed consent and authorize confidential health information to be examined in accordance with national and local subject privacy regulations.
2. The patient must have been diagnosed with clinically definite MS, at the time of informed consent.
3. The patient must be between 18-70 years of age, inclusive, at the time of informed consent.
4. The patient must have scored between 50 and 90 on the upper limb Motricity Index test, at the time of informed consent. This test evaluates strength during three essential movements (pinch grasp, elbow flexion and shoulder abduction). The selected score range criteria determine patients who suffer a moderate decline in function abilities of the upper limb.

Exclusion Criteria:

1. Onset of multiple sclerosis exacerbation within 60 days of screening.
2. History of seizures or evidence of epileptic form activity found on a screened electroencephalogram.
3. Changes in concomitant medications to avoid related changes in multiple sclerosis symptoms during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Nine-Hole Peg Test | Changes in the Nine-Hole Peg Test from Baseline to end of Second week
  The Nine-Hole Peg Test is a brief, standardized, quantitative test of upper extremity function
Nine-Hole Peg Test | Changes in the Nine-Hole Peg Test from Baseline to end of first week
  The Nine-Hole Peg Test is a brief, standardized, quantitative test of upper extremity function
Nine-Hole Peg Test | Changes in the Nine-Hole Peg Test from end of second week to follow up 2-weeks after end of intervention phase
  The Nine-Hole Peg Test is a brief, standardized, quantitative test of upper extremity function

SECONDARY OUTCOMES:
Box and Block test | Changes in the Box and Block Test from Baseline to end of Second week
  The box and blocks test (BBT) examines manual dexterity
Box and Block test | Changes in the Box and Block Test from Baseline to end of first week
  The box and blocks test (BBT) examines manual dexterity
Box and Block test | Changes in the Box and Block Test from end of second week to follow up 2-weeks after end of intervention phase
  The box and blocks test (BBT) examines manual dexterity
Isometric grip force and motor fatigue | Changes in the Isometric grip force and motor fatigue tests from baseline to end of Second week
  Peak isometric grip force (in NM) and isometric fatigue index will be determined by a hand-held dynamometer (Biometrics Ltd., USA). The hand-held dynamometer is a medical device used to assess grip strength in functional assessment and in initial and ongoing evaluation of patients with hand dysfunction
Isometric grip force and motor fatigue | Changes in the Isometric grip force and motor fatigue tests from baseline to end of first week
  Peak isometric grip force (in NM) and isometric fatigue index will be determined by a hand-held dynamometer (Biometrics Ltd.,USA). The hand-held dynamometer is a medical device used to assess grip strength in functional assessment and in initial and ongoing evaluation of patients with hand dysfunction
Isometric grip force and motor fatigue | Changes in the Isometric grip force and motor fatigue tests from end of second week to follow up 2-weeks after end of intervention phase
  Peak isometric grip force (in NM) and isometric fatigue index will be determined by a hand-held dynamometer (Biometrics Ltd.,USA). The hand-held dynamometer is a medical device used to assess grip strength in functional assessment and in initial and ongoing evaluation of patients with hand dysfunction
Sensory evaluation | Changes in the Sensory evaluation Test from Baseline to end of Second week
  The two-point discrimination test will be used to determine tactile sensation. Light-touch and pressure-sensation thresholds will be determined using monofilaments
Sensory evaluation | Changes in the Sensory evaluation Test from Baseline to end of first week
  The two-point discrimination test will be used to determine tactile sensation. Light-touch and pressure-sensation thresholds will be determined using monofilaments
Sensory evaluation | Changes in the Sensory evaluation Test from end of second week to follow up 2-weeks after end of intervention phase
  The two-point discrimination test will be used to determine tactile sensation. Light-touch and pressure-sensation thresholds will be determined using monofilaments
Patient rating scale - Disabilities of the Arm, Shoulder and Hand (DASH) | Changes in the DASH Test from Baseline to end of Second week
  The DASH (http://www.dash.iwh.on.ca/) has 30 items grouped into one scale aiming to measure 'physical function and symptoms' in people with disorders of the upper limb.15 Items are scored from 1 (no difficulty) to 5 (unable). A total 'disability/symptom' score is generated by summing items, and averaging to produce a mean item score between 1 and 5
Patient rating scale - Disabilities of the Arm, Shoulder and Hand (DASH) | Changes in the DASH Test from Baseline to end of first week
  The DASH (http://www.dash.iwh.on.ca/) has 30 items grouped into one scale aiming to measure 'physical function and symptoms' in people with disorders of the upper limb.15 Items are scored from 1 (no difficulty) to 5 (unable). A total 'disability/symptom' score is generated by summing items, and averaging to produce a mean item score between 1 and 5
Patient rating scale - Disabilities of the Arm, Shoulder and Hand (DASH) | Changes in the DASH Test from end of second week to follow up 2-weeks after end of intervention phase
  The DASH (http://www.dash.iwh.on.ca/) has 30 items grouped into one scale aiming to measure 'physical function and symptoms' in people with disorders of the upper limb.15 Items are scored from 1 (no difficulty) to 5 (unable). A total 'disability/symptom' score is generated by summing items, and averaging to produce a mean item score between 1 and 5

CONTACTS AND LOCATIONS:
Overall Officials: Anat Achiron, MD, PhD, Study Director — Multiple Sclerosis Center, Sheba Medical Hospital
Locations (1):
- Multiple Sclerosis Center, Tel Litwinsky, Ramat-gan, Israel

REFERENCES:
- [Background] Johansson S, Ytterberg C, Claesson IM, Lindberg J, Hillert J, Andersson M, Widen Holmqvist L, von Koch L. High concurrent presence of disability in multiple sclerosis. Associations with perceived health. J Neurol. 2007 Jun;254(6):767-73. doi: 10.1007/s00415-006-0431-5. Epub 2007 Apr 2. PMID 17401746
- [Background] Judge SI, Bever CT Jr. Potassium channel blockers in multiple sclerosis: neuronal Kv channels and effects of symptomatic treatment. Pharmacol Ther. 2006 Jul;111(1):224-59. doi: 10.1016/j.pharmthera.2005.10.006. Epub 2006 Feb 9. PMID 16472864
- [Background] Goodman AD, Brown TR, Krupp LB, Schapiro RT, Schwid SR, Cohen R, Marinucci LN, Blight AR; Fampridine MS-F203 Investigators. Sustained-release oral fampridine in multiple sclerosis: a randomised, double-blind, controlled trial. Lancet. 2009 Feb 28;373(9665):732-8. doi: 10.1016/S0140-6736(09)60442-6. PMID 19249634
- [Background] van Diemen HA, Polman CH, van Dongen TM, van Loenen AC, Nauta JJ, Taphoorn MJ, van Walbeek HK, Koetsier JC. The effect of 4-aminopyridine on clinical signs in multiple sclerosis: a randomized, placebo-controlled, double-blind, cross-over study. Ann Neurol. 1992 Aug;32(2):123-30. doi: 10.1002/ana.410320203. PMID 1510353
- [Background] Stefoski D, Davis FA, Fitzsimmons WE, Luskin SS, Rush J, Parkhurst GW. 4-Aminopyridine in multiple sclerosis: prolonged administration. Neurology. 1991 Sep;41(9):1344-8. doi: 10.1212/wnl.41.9.1344. PMID 1891078
- [Derived] Menascu S, Frid L, Kalron A. Sustained-release oral dalfampridine appears to have no impact on upper extremity function in people with multiple sclerosis: a randomized controlled trial. Ther Adv Neurol Disord. 2025 Feb 21;18:17562864251321696. doi: 10.1177/17562864251321696. eCollection 2025. PMID 39990866